CLINICAL TRIAL: NCT04539132
Title: Maintaining Independence and Quality of Life in Aging Adults Through Targeted Cognitive Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kwantlen Polytechnic University (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other); ABI Wellness Inc (Unknown); Watson Centre Society for Brain Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103298
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The participants will be divided into two groups (N = 20). One group will be the "intervention group" who will participate in the 6-month interdisciplinary comprehensive rehabilitation program whereas the "non-intervention" group or control group will have all of the same pre-tests administered as the intervention group, however, will not participate in the cognitive program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The "intervention group" will participate in the 6-month interdisciplinary comprehensive rehabilitation program. The ABI Wellness (ABIW) program aimed at this population would be 7 hours a week (2 days per week will be scheduled for the intervention group), consisting of around 4 hours of cognitive training (through specified drills, cognitive exercises focused on executive functioning), 1 hour of physical exercise, 1 hour of mindfulness sessions (meditation) and scheduled break times.
  Interventions: Behavioral: ABI Wellness Program
- Control Group (No Intervention): The "non-intervention" group or control group will have all the same pre-tests administered as the intervention group, however, will not participate in the cognitive program. The control group will be required to complete the assessment periods only, however, keep a record of their daily activities in a log format which is presented in the materials included herein. No other intervention or programming will be provided.

INTERVENTIONS:
Behavioral: ABI Wellness Program — The ABI Wellness program includes a computerized task which will be completed by all participants remotely. The exercise is a sustained visual-spatial processing task of progressively increasing difficulty. Subjects are presented with an analog clock face, initially showing only one hand. The subject uses a keyboard to enter a value for the hour shown. Feedback on the computer screen indicates whether the response is correct or incorrect. If the response was incorrect, the subject continues to respond until the correct response is entered. After this, a new clock face is shown. Once subjects reach a criterion of 90% accuracy over a series of consecutive responses, an additional hand is added to the clock face. Participants will complete the program at home, online, and will be required to be present on a video call during the exercise with the other participants and research assistants. The program is 150 hours over 6 months, through twice weekly 3-hour sessions.
  Arms: Intervention Group

SUMMARY:
Mild Cognitive Impairment, Alzheimer's Disease and Parkinson's Disease all represent a range of degenerative conditions that have cognitive impairments which all limit the ability for older individuals to self-manage care, participate in daily activities and community participation. The consequences of these progressive diseases increase the requirement for residential care, associated medical costs and may negatively impact the overall quality of life and mental health for individuals. According to the Alzheimer Society of Canada, over the next few decades, more than 1 million Canadian's will be living with decreased cognitive ability and will require an increased amount of support, whether through family or institutional sources.

Currently, there are few cognitive programs for individuals diagnosed with mild cognitive impairment or for individuals wishing to maintain their current level of cognitive ability which translates to meaningful improvements in daily living and independence, as well as generalized intelligence. To date, the Watson Centre Society for Brain Health (WCSBH) has successfully improved cognitive capacity, executive function and quality of life for over 100 individuals following a wide range of brain injury, and currently has a 77% return to work rate following completion of the full program. The program includes a combination of physical exercise, cognitive training and mindfulness meditation.

The purpose of the research study is to explore the impact of an interdisciplinary cognitive rehabilitation program has upon the cognitive functioning and quality of life for individuals who are assessed to have mild cognitive impairment (MCI). In particular, the aims of this study include: 1) To evaluate changes in cognition and quality life in older adults with MCI. 2) To explore the potential for intensive cognitive intervention in slowing cognitive degeneration in older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

* T-MoCA score between 19 - 23

Exclusion Criteria:

* Potential participants are under the age of 65 years at the time of screening
* Scoring results in a range outside of 19-23 on the MoCA
* Those who have have a diagnosed illness or diagnosed injury which is known to directly and negatively impact cognition
* Are known (legally) to be deemed incapable; unable to appreciate information that is relevant to making decisions or is unable to appreciate the reasonably foreseeable consequences of either making or not making a decision.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Pre-post assessment completed 6 months apart with a 6 month follow up
  Telephone Montreal Cognitive Assessment (T- MoCA) - non-invasive screening tool which takes approximately 10 minutes to complete. Thirty items assessing multiple cognitive domains are contained in the MoCa: short-term memory; visuospatial abilities via clock drawing; and a cube copy task; executive functioning via an adaptation of Trail Making phonemic fluency, and verbal abstraction; attention, concentration, and working memory via target detection, serial subtraction, digits forward, and digits backward; language via confrontation naming with low-familiarity animals, and repetition of complex sentences; and orientation to time and place (Nasreddine et al., 2005). The MoCA is scored by obtaining an item total.
Memory Alteration Test | Pre-post assessment completed 6 months apart with a 6 month follow up
  Memory Alteration Test (M@T) - A non-invasive memory screening test used to discriminate between subjects with subjective memory complaints (SMC) Without objective memory impairment and patients with amnesic mild cognitive impairment (A-MCI) and with Mild Alzheimers disease (AD). (M@T), which is a memory screening test, capable for discriminating between subjects with subjective memory complaints (SMC) (without objective memory impairment) and patients with amnestic mild cognitive impairment (A-MCI) and with mild Alzheimer's disease (AD). This is a cognitive test with high internal consistency and validity, short application (5-10 min), easy to perform and to interpret (Carnero-Pardo et al., 2011a).
Mild Cognitive Impairment Questionnaire | Pre-post assessment completed 6 months apart with a 6 month follow up
  Mild Cognitive Impairment Questionnaire (MCQ) -QOL will be measured using the 13-item MCQ tool designed to take 5 minutes to administer. The MCQ tool uses a scale of 0-4 (none, rarely, sometimes, often, or always) to assess two constructs - Practical Concerns and Emotional Concerns. Scores are transformed and presented on a metric of 0 (no problems) to 100 (maximum impact of MCI). Scale scores are interpreted using the following guide: a scale score of 0-20 indicates 'never' experiencing the issue, 21-40 'rarely' experiencing it, 41-60 'sometimes' experiencing it,61-80 'often' experiencing it, 81-100 'always' experiencing it. The MCQ has been shown to have great stability and reliability through test-retest and substantial validity with this population.
Neuro-QOL | Pre-post assessment completed 6 months apart with a 6 month follow up
  Neuro-QOL This research tool measures the physical, mental, and social effects experienced by adults with neurological conditions. The measurement takes approximately 30 minutes to complete and will be administered three times.

SECONDARY OUTCOMES:
Qualitative Interviews | Pre-post assessment completed 6 months apart with a 6 month follow up
  Interviews - Semi-structured interviews will occur with all participants in the study including the intervention and the control group with a focus upon lived experience specific to quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tess Kroeker, PhD, Principal Investigator — Kwantlen Polytechnic University; Shaun Porter, MSc, Study Director — ABI Wellness Inc

IPD SHARING:
Plan to Share IPD: No